CLINICAL TRIAL: NCT05467189
Title: Population Pharmacokinetics, Effectiveness and Safety of Antineoplastic Drugs in Elderly Patients
Brief Title: Antineoplastic Drugs in Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Qianfoshan Hospital (Other); The Second Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: Elderly-Antineoplastic drugs
Record Dates: First submitted 2022-07-04; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cancer
Keywords: Population Pharmacokinetics; Effectiveness; Safety; Antineoplastic Drugs; Elderly Patients
MeSH Terms: conditions — Neoplasms | interventions — Busulfan; Paclitaxel; Afatinib; ceritinib; Crizotinib; Antineoplastic Agents; Imatinib Mesylate; Lapatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treatment: The use of antineoplastic agents depends on the clinical practice.
  Interventions: Drug: Busulfan, Paclitaxel, Afatinib, Ceritinib, Crizotinib (Antineoplastic drugs)

INTERVENTIONS:
Drug: Busulfan, Paclitaxel, Afatinib, Ceritinib, Crizotinib (Antineoplastic drugs) — As part of routine treatment.
  Other Names: Busulfan, Paclitaxel, Afatinib, Ceritinib, Crizotinib, Imatinib, Lapatinib, etc

SUMMARY:
The purpose is to study the population pharmacokinetics, effectiveness and safety of antineoplastic drugs (Busulfan, Paclitaxel, Afatinib, Ceritinib, Crizotinib, Imatinib, Lapatinib, etc) in elderly patients and recommend optimized dosage regimens.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in the study:

1. Age ≥65 years old;
2. Diagnosed with cancer;
3. Using antineoplastic drugs for treatment.

Exclusion Criteria:

Subjects with any of the following criteria will not be enrolled in this study:

1. Patients who are expected to die within 48 hours;
2. Patients with allergy to antineoplastic drugs;
3. Patients receiving other investigational drugs;
4. Other factors that the researcher considers unsuitable for inclusion.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with cancer (≥65years)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The peak plasma drug concentration of antineoplastic drugs. | at (0-4) hours after administration
  To detect the peak plasma drug concentration of antineoplastic drugs.
The random plasma drug concentration of antineoplastic drugs. | at (4-10) hours after administration
  To detect the random plasma drug concentration of antineoplastic drugs.
The trough plasma drug concentration of antineoplastic drugs. | at (1-2) hours before the next administration
  To detect the trough plasma drug concentration of antineoplastic drugs.

SECONDARY OUTCOMES:
Objective ResponseRate ,ORR | Enrollment to end of treatment up to 5 years
Overall Survival ,OS | First day of study treatment to the date of death due to any cause, assessed up to 5 years
Progression-free Survival ,PFS | First day of study treatment to the date of disease progression or death due to any cause, assessed up to 5 years
Time to Progression ,TTP | Enrollment to end of treatment up to 5 years
The incidence of adverse drug reaction | Enrollment to end of treatment up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wei, Ph.D, Study Chair — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China